CLINICAL TRIAL: NCT02500836
Title: Phase III Topical Application of Cocaine HCl 4% Solution on Safety/Efficacy & Cocaine HCl 4% & 10% Solution on Safety in Local Anesthesia for Diagnostic Procedures & Surgeries on or Through Accessible Mucous Membranes of the Nasal Cavities
Brief Title: Topical Application of Cocaine HCl 4%, or 10%, or Placebo Solution in Local (Topical) Anesthesia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lannett Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COCA4vs10-002
Record Dates: First submitted 2015-07-12; First posted 2015-07-17 (Estimated); Results first posted 2017-05-16 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-04

CONDITIONS: Any Ear Nose or Throat Conditions; With Identified Need for a Diagnostic Procedure or Surgery on or Through the Mucous Membranes of the Nasal Cavities
Keywords: Ear; Nose; Throat
MeSH Terms: interventions — Cocaine; Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cocaine HCI 4% Topical Solution (Experimental): Cocaine HCl 4% Topical Solution, up to 4 mL, is applied for 20 minutes via cotton or rayon pledget(s), then the nasal site is tested with a Von Frey (or equivalent) filament (Size 5.88, about 60 grams of force) to determine and record whether the subject has a pain score of 0 (zero) (0 = No Pain, 10 = Unbearable pain) after treatment application compared to the Von Frey filament test right before treatment application. If a pain score of 0 (zero) is recorded, then the diagnostic procedure or surgery proceeds along with safety monitoring for at least 90 minutes after removal of the pledget(s). The subject will be followed for safety for seven days. The total number of pledgets used, and the amount of Cocaine HCl 4% topical solution used (1 mL per pledget) will be recorded.
  Interventions: Drug: Cocaine HCl 4% Topical Solution
- Cocaine HCI 10% Topical Solution (Experimental): Cocaine HCl 10% Topical Solution, up to 4 mL, is applied for 20 minutes via cotton or rayon pledget(s), then the nasal site is tested with a Von Frey (or equivalent) filament (Size 5.88, about 60 grams of force) to determine and record whether the subject has a pain score of 0 (zero) (0 = No Pain, 10 = Unbearable pain) after treatment application compared to the Von Frey filament test right before treatment application. If a pain score of 0 (zero) is recorded the application then proceed with the diagnostic procedure or surgery along with safety monitoring for at least 90 minutes post removal of pledgets, and, the subject will be followed for safety for at least seven days post solution application. The total number of pledgets used, and the amount of Cocaine HCl 10% topical solution used (1 mL per pledget) will be recorded.
  Interventions: Drug: Cocaine HCl 10% Topical Solution
- Placebo Topical Solution (Placebo Comparator): Placebo Topical Solution, up to 4 mL, is applied for 20 minutes via cotton or rayon pledget(s), then the nasal site is tested with a Von Frey (or equivalent) filament (Size 5.88, about 60 grams of force) to determine and record whether the subject has a pain score of 0 (zero) (0 = No Pain, 10 = Unbearable pain) after treatment application compared to the Von Frey filament test right before treatment application. The subject will then exit the treatment portion of the trial and be followed for safety for seven days . The total number of pledgets used, and the amount of placebo solution used (1 mL per pledget) will be recorded. After a minimum of 90 minutes from the time of study drug pledget removal, the subjects may have their surgery or diagnostic procedure, and the treatment reverts to standard anesthetic management (e.g. application of lidocaine, tetracaine, bupivicaine or other suitable products at the discretion of the investigator).
  Interventions: Drug: Placebo Topical Solution

INTERVENTIONS:
Drug: Cocaine HCl 4% Topical Solution — Topical solution, up to 4 mL, is applied for 20 minutes via cotton or rayon pledget(s) to the accessible mucous membranes of the nasal cavities.
  Arms: Cocaine HCI 4% Topical Solution
Drug: Cocaine HCl 10% Topical Solution — Topical solution, up to 4 mL, is applied for 20 minutes via cotton or rayon pledget(s) to the accessible mucous membranes of the nasal cavities.
  Arms: Cocaine HCI 10% Topical Solution
Drug: Placebo Topical Solution — Topical solution, up to 4 mL, is applied for 20 minutes via cotton or rayon pledget(s) to the accessible mucous membranes of the nasal cavities.
  Arms: Placebo Topical Solution

SUMMARY:
Randomized, prospective, multi-center, double blind placebo-controlled parallel group study of a Placebo Topical Solution versus Cocaine HCl 4% Topical Solution for safety and efficacy, and Cocaine HCl 4% and 10% Topical Solution for Safety as an anesthetic prior to a diagnostic procedure or surgery on or through accessible mucous membranes of the nasal cavities. Both domestic (United States) and foreign sites are eligible, and both inpatient and outpatient settings are eligible.

DETAILED DESCRIPTION:
Eligible subjects will undergo either an office-based or operating room-based procedure or surgery. The approximately 620 subjects will be randomized in a 2:2:1 fashion to one of the three treatment groups (248 subjects randomized to the Cocaine HCl 4% solution, 248 subjects randomized to the Cocaine HCl 10%, and 124 subjects randomized to the placebo solution) pre-procedure and given one application of the assigned test product with Von Frey filament testing occurring after application.

ELIGIBILITY:
Inclusion Criteria:

- Subjects must meet all of the following criteria prior to enrollment in the study:

* Provide written informed consent and HIPAA authorization. Residents of California must also review and sign the California Subject Bill of Rights.
* Male or female ≥18 years of age.
* Predetermined need from a physician for diagnostic procedure or surgery on or through the nasal mucous membranes of either one or two nostrils that merits the use of anesthesia.
* Ability to feel pain sensation normally in the nasal mucous membranes, as verified via Von Frey 5.88 monofilament testing
* Ability to clearly communicate pain and sensation of the nasal mucous membranes.

Exclusion Criteria:

* Has a known allergy to any ester based anesthetics including cocaine, procaine, tetracaine, chlorprocaine, dibucaine, or benzocaine and/or any other compounds of the drugs and/or devices that are part of this protocol. (Amide based or other non-ester based anesthetic allergies are NOT exclusionary. Amide based anesthetics are: Lidocaine, Mepivicaine, Bupivicaine, Levobupivicaine, Ropivicaine, Etidocaine, Prolicaine, and Articaine).
* Has a history of abuse of controlled substances, nasal or otherwise, or has damage to the nasal space, that in the opinion of the investigator might interfere with the ability of the subject or the investigator to judge anesthesia from the trial drug.
* Has used any investigational drug(s) within 30 days preceding the randomization.
* Is pregnant or is a nursing mother
* Women of childbearing potential (WOCBP) and male partners of WOCBP who are not willing to use an acceptable method of contraception to avoid pregnancy throughout the study. Contraceptive practices must extend for women at least 30 days and for male partners of WOCBP at least 90 days after the last dose of investigational product in such a manner that the risk of pregnancy or risk to a pregnancy is minimized.
* Is < 18 years of age
* Suffers from a condition, other than the need for a diagnostic procedure or surgery on or through the nasal mucous membranes which, in the opinion of the Investigator, would compromise the safety of the subject, the quality of the data, or the normal wound healing process.
* Use of any analgesic 2 days prior to screening or has a need to use these drugs during the screening period. This includes NSAIDs, such as ibuprofen, diclofenac, indomethacin, sulindac, tolmetin, ketoprofen, flurbiprofen, naproxen, opioids such as codeine, hydrocodone, hydromorphone, morphine, oxycodone, aspirin, or acetaminophen.
* Subjects who have experienced a seizure while taking isoniazid (INH), phenothiazines, chlorpromazine, thioridazine, theophylline, or tricyclic antidepressants such as amitriptyline.
* Has previously received study drug during this study. Subjects who fail screening may rescreen if eligibility requirements are met, but only if the subject has not received any study drug during this study.
* Has a history of myocardial infarction, coronary artery disease, congestive heart failure, irregular heart rhythm (as fully defined in sections 7.9.4, 7.9.5 and 7.9.6) or uncontrolled hypertension or is taking monoamine oxidase inhibitors (6). Uncontrolled hypertension is defined as systolic blood pressure greater than or equal to 140 mm Hg or diastolic blood pressure greater than or equal to 90 mm Hg (43)(44).
* Has a known personal or family history of hereditary pseudocholinesterase deficiency. (2) Study participants will be screened by asking about personal or family history of anesthetic reaction, anesthetic death, and previous diagnosis of pseudocholinesterase deficiency in a relative or personally. Subjects identified with pseudocholinesterase deficiency are at risk for delayed recovery with certain anesthetics (e.g. succinylcholine and ester-based anesthetics). (14)
* Has a known personal or family history of pheochromocytoma. (2) Study participants will be specifically asked if they have been treated for a pheochromocytoma previously or if they have a family member who has been diagnosed with pheochromocytoma (since 10% of these are familial). (14)
* Has a known personal or family history of an adrenal tumor.
* Use of amphetamines in the 2 days prior to screening or has a need to use these drugs during the course of the study. All stimulant prescription, and nonprescription products such as catecholamines (norepinephrine or epinephrine), ephedrine, pseudoephedrine and any other amphetamines in the 48 hours prior to screening or has a need to use these drugs during the course of the study. All herbal products except coffee, tea, or herbal tea are also prohibited within 48 hours prior to screening or if the subject has a need to use these drugs during the course of the study. Coffee, Tea, and Herbal Tea are not exclusionary criteria or prohibited medications as they are food products not prescription or nonprescription products.
* Has screening 12-lead ECG findings of any abnormalities as listed in section 7.9.4, 7.9.5, and 7.9.6. Generally, these are current or prior myocardial ischemia or infarction, dysrhythmia, or risk of serious dysrhythmia (such as prolonged QT interval) and include any other clinically significant abnormal ECG finding that, in the opinion of the Investigator in consultation with the Medical Monitor, may potentially result in this trial being unsafe for the subject.
* An exception to this would be 7.9.5.11 (resting sinus bradycardia or resting sinus tachycardia to a limit of 110 beats per minute) as these represent normal variants that may be found in younger or older healthy adults. (36)
* Hemoglobin <8.5 g/dL; a one-time retest will be allowed for Hb 8.3- 8.4 g/dL
* WBC < 3.5 x 103 cells/mcL; a one-time retest will be allowed for WBC 3.3-3.4 x 103 cells/mcL
* Platelets < 100 x 103 platelets/mcL; a one-time retest will be allowed for platelets 90-99x 103 platelets/mcL
* Serum Potassium <3.5 or >5.0 mEq/L
* Serum ALT, AST, and bilirubin exceeding 2X ULN for the lab's reference values
* Cardiac enzymes above the range of normal
* Coagulation studies that in the opinion of the investigator would be cause for the subject to be excluded from the study.
* Positive urine pregnancy test at screening or Day 1
* Positive urine drug test at screening or Day 1 without prior medically-necessary use of controlled substances (for example, benzodiazepines for anxiety)
* Subjects is a member of the Investigational Team, including Investigators or Sub-Investigators, or their immediate family.

A one-time retest is permitted for any blood test if the original sample was hemolyzed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 646 (Actual)
Dates: Start 2015-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Richmond ENT, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from patients scheduled for an office-based or operating room-based diagnostic procedure or surgery on or through accessible mucous membranes of the nasal cavities.
Pre-assignment Details: A screening visit was conducted to ensure that each subject met inclusion/exclusion criteria for the study. Subjects who met all eligibility criteria were then enrolled for the drug application and procedure visit, which may have been on the same day as the screening visit.
Groups:
- Cocaine HCI 4% Topical Solution: Subjects randomized to receive Cocaine HCl 4% Topical Solution
- Cocaine HCI 10% Topical Solution: Subjects randomized to receive Cocaine HCl 10% Topical Solution
- Placebo Topical Solution: Subjects randomized to receive Placebo Topical Solution
Period: Overall Study
Arm/Group | Cocaine HCI 4% Topical Solution | Cocaine HCI 10% Topical Solution | Placebo Topical Solution
Started | 259 | 259 | 128
Completed | 256 | 254 | 127
Not Completed | 3 | 5 | 1

BASELINE CHARACTERISTICS:
Population: The analysis of baseline characteristics includes all enrolled subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cocaine HCI 4% Topical Solution | Cocaine HCI 10% Topical Solution | Placebo Topical Solution | Total
Number analyzed (Participants) | 259 | 259 | 128 | 646
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.42 (13.34) | 37.50 (12.76) | 36.01 (12.34) | 37.57 (12.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 169 | 156 | 68 | 393
  Male | 90 | 103 | 60 | 253
Region of Enrollment [Number; unit: participants]
  United States | 259 | 259 | 128 | 646

OUTCOME MEASURES:

1. Primary Outcome: Immediate and Sustained Anesthetic Success for Cocaine HCl 4% Topical Solution and Placebo Topical Solution
Description: Subjects who meet the following for each nostril that received the study drug application are considered a treatment success: Prior to the diagnostic procedure or surgery, based on the von Frey monofilament test, after application of the assigned study drug solution (Cocaine HCl 4% Topical Solution or Placebo Topical Solution), the subject response is a 0 (zero) pain score on the 11 point pain scale (0 = no pain, 10 = unbearable pain) compared to the von Frey monofilament test right before study drug application. And, during the diagnostic procedure or surgery, no further analgesic treatment is required (only 4% Cocaine HCl subjects who receive a diagnostic procedure or surgery). Subjects with missing primary outcome data are marked as treatment failures in both treatment groups.
Time Frame: One Day, Single office based diagnostic procedure or surgery
Population: The analysis of primary outcome data is based on an intent-to-treat population, which includes all randomized subjects who received study drug.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cocaine HCI 4% Topical Solution | Placebo Topical Solution
Number analyzed (Participants) | 258 | 127
proportion of participants | 0.7093 [0.6498 to 0.7640] | 0.1969 [0.1316 to 0.2767]
Statistical Analysis 1: Comparison: Cocaine HCI 4% Topical Solution vs Placebo Topical Solution; The null hypothesis is that the proportions of treatment group successes are equal; Test type: Superiority; p < 0.0001, Fisher Exact — One-sided p-value

2. Secondary Outcome: Immediate and Sustained Anesthetic Success for Cocaine HCl 10% Topical Solution
Description: Subjects who meet the following for each nostril that received the study drug application are considered a treatment success: Prior to the diagnostic procedure or surgery, based on the von Frey monofilament test, after application of the assigned study drug solution (Cocaine HCl 10% Topical Solution), the subject response is a 0 (zero) pain score on the 11 point pain scale (0 = no pain, 10 = unbearable pain) compared to the von Frey monofilament test right before study drug application. And, during the diagnostic procedure or surgery, no further analgesic treatment is required (only 10% Cocaine HCl subjects who receive a diagnostic procedure or surgery).
Time Frame: One Day, Single office based diagnostic procedure or surgery
Population: The analysis of secondary outcome data is based on an intent-to-treat population, which includes all randomized subjects who received study drug. The analysis of this secondary efficacy endpoint includes comparisons to the primary endpoint for the Placebo Topical Solution treatment group.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cocaine HCI 10% Topical Solution | Placebo Topical Solution
Number analyzed (Participants) | 254 | 127
proportion of participants | 0.8268 [0.7745 to 0.8712] | 0.1969 [0.1316 to 0.2767]
Statistical Analysis 1: Comparison: Cocaine HCI 10% Topical Solution vs Placebo Topical Solution; The null hypothesis is that the proportions of treatment group successes are equal; Test type: Superiority; p < 0.0001, Fisher Exact — One-sided p-value

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for each subject from the time informed consent was signed until termination from the study.
Arm/Group | Cocaine HCI 4% Topical Solution | Cocaine HCI 10% Topical Solution | Placebo Topical Solution
Serious Adverse Events (participants affected / at risk) | 0/259 | 0/259 | 0/128
Other Adverse Events (participants affected / at risk) | 218/259 | 237/259 | 94/128
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cocaine HCI 4% Topical Solution (N=259) | Cocaine HCI 10% Topical Solution (N=259) | Placebo Topical Solution (N=128)
Atrioventricular Block First Degree (Cardiac disorders) | 1 | 2 | 3
Bradycardia (Cardiac disorders) | 8 | 1 | 5
Sinus Tachycardia (Cardiac disorders) | 6 | 9 | 0
Tachycardia (Cardiac disorders) | 12 | 28 | 1
Tachycardia Paroxysmal (Cardiac disorders) | 2 | 6 | 1
Nausea (Gastrointestinal disorders) | 3 | 3 | 0
Electrocardiogram QRS Complex Prolonged (Investigations) | 4 | 8 | 3
Electrocardiogram QT Prolonged (Investigations) | 7 | 10 | 3
Heart Rate Increased (Investigations) | 2 | 7 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 8 | 0
Dizziness (Nervous system disorders) | 2 | 3 | 0
Headache (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0
Anxiety (Psychiatric disorders) | 4 | 0 | 0
Nasal Septum Deviation (Respiratory, thoracic and mediastinal disorders) | 11 | 16 | 2
Nasal Turbinate Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 3
Diastolic Hypertension (Vascular disorders) | 2 | 4 | 1
Hypertension (Vascular disorders) | 201 | 220 | 85
Hypotension (Vascular disorders) | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor right of review of publication, right to remove confidential or proprietary information, and all multi-center data publication done before any additional publications.